CLINICAL TRIAL: NCT05658497
Title: Vumerity (Diroximel Fumarate) Prospective MS Pregnancy Exposure Registry
Brief Title: Pregnancy Exposure Registry for Vumerity (Diroximel Fumarate)
Status: Recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 272MS401
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Pregnancy; Relapsing forms of MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — diroximel fumarate; Interferon beta-1a; Natalizumab; Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Diroximel Fumarate: Pregnant women with MS who were exposed to DRF at any time from 2 weeks after the first day of their LMP through the end of pregnancy.
  Interventions: Drug: Diroximel Fumarate
- Disease Modifying Therapy (DMTs) Exposed: Pregnant women with MS who were exposed to other DMTs (e.g., Avonex and Tysabri Pregnancy Registries) at any time from 2 weeks after the first day of their LMP through the end of pregnancy.
  Interventions: Drug: Avonex; Biological: Tysabri
- DMTs Unexposed: Pregnant women who were unexposed to DMT which is defined as either never received a DMT or discontinued treatment with DRF at least 1 day before 2 weeks after the first day of their LMP or discontinued a non-Registry-specified MS DMT more than 5 times its half-life prior to 2 weeks after the first day of their LMP.
- Dimethyl Fumarate: Pregnant women with MS who were exposed to DMF at any time from 2 weeks after the first day of their LMP through the end of pregnancy.
  Interventions: Drug: Dimethyl Fumarate
- Women Without MS: Pregnant women with external, general population comparators.

INTERVENTIONS:
Drug: Diroximel Fumarate — Administered as specified in the treatment arm.
  Other Names: VUMERITY; BIIB098
  Groups: Diroximel Fumarate
Drug: Avonex — Administered as specified in the treatment arm.
  Other Names: BG9418; interferon beta-1a
  Groups: Disease Modifying Therapy (DMTs) Exposed
Biological: Tysabri — Administered as specified in the treatment arm.
  Other Names: Natalizumab; BG00002
  Groups: Disease Modifying Therapy (DMTs) Exposed
Drug: Dimethyl Fumarate — Administered as specified in the treatment arm.
  Other Names: Tecfidera; DMF; BG00012
  Groups: Dimethyl Fumarate

SUMMARY:
The primary objectives of the study are to estimate the risk of major congenital malformations (MCMs) in infants born to women with multiple sclerosis (MS) who were exposed to diroximel fumarate (DRF) at any time from 2 weeks after the first day of their last menstrual period (LMP) up through the first trimester of pregnancy and to comparatively evaluate pregnancy outcomes with MCMs in women with MS who were exposed to DRF at any time from 2 weeks after the first day of their LMP through the first trimester of pregnancy with the following: i) women with MS who were unexposed to disease modifying therapies (DMTs) and, ii) women with MS who were exposed to other DMTs (e.g., Avonex and Tysabri Pregnancy Registries).

The secondary objective of the study is to evaluate pregnancy outcomes in women with DRF exposure at any time from 2 weeks after the first day of their LMP through the end of pregnancy compared with the following: i) women with MS who were unexposed to DMTs, ii) women with dimethyl fumarate (DMF) exposure, iii) women with MS who were exposed to other DMTs (e.g., Avonex and Tysabri Pregnancy Registries), and iv) women without MS (e.g., women from external, general population comparators).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have a diagnosis of MS
* Documentation that the participant was one of the following:

  1. exposed to DRF at any time from 2 weeks after the first day of their LMP (i.e., conception date) up through any time during pregnancy. (If exact exposure dates are unknown, the reporter must be able to specify or estimate trimester of exposure).
  2. unexposed to any DMT during pregnancy, defined as having never received DMT therapy; discontinued treatment with DRF at least 1 day before 2 weeks after the first day of their LMP (i.e., conception date); or discontinued a non Registry-specified MS DMT more than 5 times its half-life prior to 2 weeks after the first day of their LMP (i.e., conception date)
* Participants with knowledge of the outcome of the pregnancy (e.g., pregnancy loss or live birth)

Key Exclusion Criteria:

- None

NOTE: Other protocol defined Inclusion criteria may apply

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will include pregnant female participants with MS who were exposed to DRF at any time from 2 weeks after the first day of their LMP up through any time during pregnancy and compared with pregnancies among women with MS who were exposed to DMF, women with MS who were exposed to other DMTs (e.g., Avonex and Tysabri Pregnancy Registries), women with MS who were unexposed to DMTs, and women without MS.
  Participants will be classified into 2 enrolment types, Prospective and Retrospective. Prospective registration:a report of a pregnancy enrolled prior to knowledge of the pregnancy outcome, including prior to the detection of a congenital malformation at prenatal testing. Women who enrol after any knowledge of the pregnancy outcome will be enrolled as retrospective cases but will not be included in the primary analysis, i.e.,pregnancies with a prenatal testing result indicative of any congenital malformation/pregnancies with known outcomes at time of initial report.
Sampling Method: Non-Probability Sample
Enrollment: 908 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2032-07-06 (Estimated); Study Completion 2032-07-06 (Estimated)

PRIMARY OUTCOMES:
Number of Major Congenital Malformations (MCMs) | Up to 52 weeks postdelivery
  MCMs include abnormalities in structural development that are medically or cosmetically significant are present at birth, and persist in postnatal life unless or until repaired as evaluated by independent advisors used throughout the registry.

SECONDARY OUTCOMES:
Number of Elective or Therapeutic Terminations | Up to 9 months of pregnancy
  Elective or therapeutic pregnancy termination is any induced or voluntary fetal loss during pregnancy. It will be subclassified as elective or therapeutic pregnancy terminations as whether it was due to a fatal anomaly or not.
Number of Spontaneous Abortions | Before 22 weeks of gestation
  Spontaneous abortion is defined as any loss of a fetus due to natural causes before 22 weeks of gestation.
Number of Fetal Deaths Including Still Birth | At or after 22 weeks of gestation
  Fetal death or stillbirth refers to the death of a fetus prior to complete expulsion or extraction from its mother at or after 22 weeks of gestation. Death is indicated by the fact that, after such separation, the fetus does not show any evidence of life (e.g., heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles). Fetal death occurring at or after 22 weeks but before 28 weeks of gestation is considered an early fetal loss. Fetal death occurring at or after 28 weeks is considered a late fetal loss.
Number of Live Births | Up to delivery (approximately 10 months)
  A live birth refers to a complete expulsion or extraction from its mother of a surviving neonate breathing, or showing any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles, whether the umbilical cord has been cut or the placenta is attached. Any live birth before 37 weeks of gestation will be considered premature birth. Any live birth at or after 37 weeks but before 42 weeks of gestation will be considered full-term birth. Any live birth at or after 42 weeks of gestation will be considered post-term birth.
Number of Ectopic Pregnancies | Up to 9 months of pregnancy
Number of Molar Pregnancies | Up to 9 months of pregnancy
Number of Maternal Deaths | Up to 12 weeks postdelivery
  Maternal death is death of a pregnant woman during pregnancy, labor, or delivery. Registry will also report maternal deaths that occur up to 12 weeks postdelivery.
Number of Neonatal Deaths | Prior to 28 days postdelivery
  Neonatal death is death occurring in a neonate prior to 28 days of life.
Number of Perinatal Deaths | At or after 28 days to 12 weeks postdelivery
  Perinatal death is death occurring at or after 28 days of life and prior to 12 weeks of life.
Number of Infant Deaths | Between 12 to 52 weeks postdelivery
  Infant death is death occurring between 12 and 52 weeks of life, inclusive.
Number of Serious or Opportunistic Infections in Liveborn Children | Up to 52 weeks postdelivery
Number of Infants with Abnormal Postnatal Growth and Development | Up to 52 weeks postdelivery
  Infant growth measurements will be used to estimate gender-specific weight-for-length, head circumference-for-age, length-for-age, and weight-for-age percentiles. Developmental milestones (i.e., social/emotional, language/communication, neurocognitive, movement/physical development) will be used to determine results of infant status (i.e., below, above, or at age-appropriate achievement).
Number of Participants with Pregnancy Complications | Up to 9 months of pregnancy
  Pregnancy complications may include incidences of pre-eclampsia, eclampsia, pregnancy-induced hypertension, preterm labor, gestational diabetes and placenta previa.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (7):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - IQVIA US Office, Durham, North Carolina
- Austin Hospital, Heidelberg, Australia
- Katholisches Klinikum Bochum, Bochum, North Rhine-Westphalia, Germany
- St Vincent's University Hospital, Dublin, Ireland
- Hospital Universitario Ramon y Cajal, Madrid, Spain
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/